CLINICAL TRIAL: NCT00190840
Title: Open-Label Single-Arm Phase 2 Study of ALIMTA in Patients With Advanced Non-Small Cell Lung Cancer Who Have Had Prior Chemotherapy
Brief Title: A Single Arm Phase 2 Study of Pemetrexed as 2nd-Line Treatment of Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6685; H3E-AA-S037
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

INTERVENTIONS:
Drug: pemetrexed

SUMMARY:
In previous phase 2 studies, pemetrexed has shown antitumor activity in advanced non-small cell lung cancer as a single agent as well as in combination with cisplatin. Since the introduction of vitamin supplementation, pemetrexed has shown good tolerance and high safety. Vitamin supplementation has opened the opportunity to offer patients higher pemetrexed dosing, as has been demonstrated by a recent Phase 1 study. The higher dose with supplementation may increase pemetrexed's efficacy without unduly compromising safety. The present Phase 2 study will use pemetrexed dosing that is tailored to individual patient tolerance, and is an effort to determine the efficacy and safety of this approach in patients with advanced NSCLC who had prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of NSCLC
* Locally advanced or metastatic disease (Stage IIIB or IV).
* Patients must have previously received one chemotherapy regimen for palliative therapy of locally advanced or metastatic disease.
* Disease status must be that of measurable disease as defined by RECIST criteria
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale; and adequate organ function.

Exclusion Criteria:

* Known or suspected brain metastasis, or Second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Concurrent administration of any other tumor therapy.
* History of significant neurological or mental disorder, including seizures or dementia; or any other serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed.
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186
Dates: Start 2003-09; Study Completion 2005-10

PRIMARY OUTCOMES:
Response rate according to RECIST criteria

SECONDARY OUTCOMES:
To assess the following time to event efficacy variables:
o Duration of overall response for responding patients
o Time to progressive disease
o Time to treatment failure
o Survival
To characterize the quantitative and qualitative toxicity of pemetrexed when used at tailored dosing in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chermside, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashford, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fitzroy, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hong Kong, China
- Egypt (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairo
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabad, Andhra Pradesh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludhiana, Punjab
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chandigarh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delhi
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea, Bihor County
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova, Dolj
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si, Gyeonggi-do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei, Taiwan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eskişehir, Turkey (Türkiye)